CLINICAL TRIAL: NCT05560802
Title: Can the Use of a Next Generation Partograph Based on WHO's Latest Intrapartum Care Recommendations Improve Neonatal Outcomes? a Stepped-wedge Cluster Randomized Trial (PICRINO)
Brief Title: Can the Use of a Next Generation Partograph Improve Neonatal Outcomes? (PICRINO)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Marie Blomberg, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Picrino2022
Record Dates: First submitted 2022-09-17; First posted 2022-09-29 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Neonatal Complication; Labor (Obstetrics)--Complications
Keywords: neonatal outcomes; obstetric outcomes; labour care guide

STUDY DESIGN:
Intervention Model Description: multicenter, stepped-wedge cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Labour care guide (Experimental): According to WHO guidelines
  Interventions: Other: WHOs Labour care guide
- Standard care (No Intervention): Standard delivery care in Sweden

INTERVENTIONS:
Other: WHOs Labour care guide — Guidelines for monitoring labor progress, the WHOs LCG
  Arms: Labour care guide

SUMMARY:
The overall aim is to evaluate the impact of the use of two different guidelines for monitoring labor progress, the WHOs LCG versus standard care, on neonatal and maternal outcomes. The hypothesis is that the use of LCG will reduce adverse neonatal outcomes and decrease the number of intrapartum Cesarean sections compared with standard care.

Secondly, other perinatal interventions and complications will be compared between the LCG and standard care groups, as well as economic considerations. This will be investigated using a multicenter, stepped-wedge cluster randomized trial design.

In addition, the project will explore a series of quantitative and qualitative research questions to gain in-depth knowledge about experiences and perceptions about childbirth and the use of LCG. These research questions will be investigated using questionnaires, focus group and individual interviews with providers, partners and women that have gone through childbirth.

DETAILED DESCRIPTION:
Study Title

Can the use of a next generation partograph based on WHO's latest intrapartum care recommendations improve neonatal outcomes? A stepped-wedge cluster randomized trial (PICRINO).

Primary Objectives

To compare two different guidelines for monitoring labor progress, the the World Health Organization (WHO)'s Labour Care Guide (LCG) with standard care, and evaluate:

Adverse neonatal outcome, a composite outcome of perinatal mortality and neonatal morbidity. Neonatal morbidity will include five-minute Apgar score <7, hypoxic ischemic encephalopathy II-III, intracranial hemorrhage, neonatal seizures, meconium aspiration syndrome, and admission to a neonatal unit.

The rate of intrapartum cesarean section.

Secondary Objectives

Secondary outcomes will be a composite of severe neonatal outcomes including five-minute Apgar score <4, hypoxic ischemic encephalopathy II-III, intracranial hemorrhage, neonatal seizures and meconium aspiration syndrome and other relevant neonatal outcomes.

Obstetric outcomes will be mode of delivery, oxytocin use, postpartum hemorrhage, perineal laceration (grade II-IV), duration of labor, women´s and partner´s experiences of childbirth, healthcare providers experiences of and compliance to LCG and economic considerations.

Study Design

A multicenter, stepped-wedge cluster randomized trial.

Study Population

All women in active labor at participating delivery units in Sweden.

Power analysis

With significance level 0.05, the power to detect the anticipated risk reduction (20%) would be >0.999.

Study Duration

2023-2025

ELIGIBILITY:
Inclusion Criteria:

-All women in active labor

Exclusion Criteria:

-No exclusion criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120000 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Adverse neonatal outcome | 12 weeks up to 18 months
  a composite outcome of perinatal mortality and neonatal morbidity. Neonatal morbidity will include five-minute Apgar score <7, hypoxic ischemic encephalopathy II-III, intracranial hemorrhage, neonatal seizures, meconium aspiration syndrome, and admission to a neonatal unit.
The rate of intrapartum cesarean section | 12 weeks up to 18 months
  The rate of intrapartum cesarean section

SECONDARY OUTCOMES:
Neonatal outcomes | 12 weeks up to 18 months
  Five-minute Apgar score <7
  admission to neonatal unit
  Hypoxic ischemic encephalopathy II-III
  Intracranial hemorrhage
  Neonatal seizures
  Meconium aspiration syndrome
  Five-minute Apgar score <4
  Perinatal mortality
  neonatal mortality
  Neonatal infection
  Neonatal hypoglycemia
  Neonatal jaundice
  Shoulder dystocia
  Obstetric brachial plexus injury
Obstetric outcomes | 12 weeks up to 18 months
  Rates of spontaneous vaginal delivery
  Rates of instrumental delivery
  Indications for intrapartum cesarean section
  Rates of oxytocin use for augmentation of labor
  Cervical dilation at onset of augmentation (centimeters)
  Rates of adherence to oxytocin use recommendations
  Rates of epidural use
  Amount of postpartum bleeding, ml
  Rates of perineal laceration (grade II-IV)
  Duration of labor, minutes
Childbirth experience (women and partners) | 12 weeks up to 18 months
  interviews questionaries
Provider experience of LCG | 12 weeks up to 18 months
  interviews
Economic evaluation | 12 weeks up to 18 months
  Data on health care utilization for women Data on health care utilization for children

CONTACTS AND LOCATIONS:
Overall Officials: Marie Blomberg, Professor, Principal Investigator — Department of Biomedical and Clinical Sciences, Linköping University, Linköping, Sweden.
Locations (24):
- Sweden (24):
  - Eksjö höglandssjukhuset, Eksjö
  - Falu Lasarett, Falun
  - Gällivare sjukhus, Gällivare
  - Göteborg Salgrenska Universitetssjukhuset, Gothenburg
  - Helsingborgs lasarett, Helsingborg
  - Huddinge Karolinska universitetssjukhus, Huddinge
  - Hudiksvalls sjukhus, Hudiksvall
  - Jönköping Länssjukhuset Ryhov, Jönköping
  - Länssjukhuset, Kalmar
  - Kristianstad centralsjukhus, Kristianstad
  - Linköpings universitetssjukhus, Linköping
  - Lund Skånes universitetssjukhus, Lund
  - Skellefteå Lasarett, Skellefteå
  - Södertälje Sjukhus, Södertälje
  - Sunderby sjukhus, Södra Sunderbyn
  - BB Stockholm, Stockholm
  - Stockholm Södersjukhuset, Stockholm
  - Umeå Norrlands universitetssjukhus, Umeå
  - Akademiska sjukhuset, Uppsala
  - Värnamo sjukhus, Värnamo
  - Västerviks sjukhus, Västervik
  - Visby Lasarett, Visby
  - Ystad Lasarett, Ystad
  - Vrinnevisjukhuset, Norrköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No
At present we are not allowed to share anonymized data extracted from Swedish medical health registers

REFERENCES:
- [Background] WHO recommendations: Intrapartum care for a positive childbirth experience. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK513809/ PMID 30070803
- [Background] Vogel JP, Comrie-Thomson L, Pingray V, Gadama L, Galadanci H, Goudar S, Laisser R, Lavender T, Lissauer D, Misra S, Pujar Y, Qureshi ZP, Amole T, Berrueta M, Dankishiya F, Gwako G, Homer CSE, Jobanputra J, Meja S, Nigri C, Mohaptra V, Osoti A, Roberti J, Solomon D, Suleiman M, Robbers G, Sutherland S, Vernekar S, Althabe F, Bonet M, Oladapo OT. Usability, acceptability, and feasibility of the World Health Organization Labour Care Guide: A mixed-methods, multicountry evaluation. Birth. 2021 Mar;48(1):66-75. doi: 10.1111/birt.12511. Epub 2020 Nov 22. PMID 33225484
- [Derived] Isgren AR, Korsoski R, Abrahamsson T, Wendel SB, Kallen K, Lundborg L, Remaeus K, Thomas K, Wikstrom AK, Carlsson Y, Blomberg M. Can the use of a next generation partograph based on WHO's latest intrapartum care recommendations improve neonatal outcomes? (PICRINO) Study protocol for a stepped-wedge cluster randomized trial. PLoS One. 2025 Mar 4;20(3):e0316336. doi: 10.1371/journal.pone.0316336. eCollection 2025. PMID 40036215